CLINICAL TRIAL: NCT06768541
Title: Short Stem Total Hip Arthroplasty in Patients With DORR Type C Femur Configuration: Measured Subsidence
Brief Title: Subsidence of Short Stem THA With DORR Type C
Status: Active, not recruiting | Type: Observational
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Other Study IDs: EK1330/2022
Record Dates: First submitted 2024-12-01; First posted 2025-01-10 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hip Osteoarthritis; Short Stem Prosthesis; Total Hip Arthroplasty (THA)
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dorr C Hip: Patients who received short stem THA with a Dorr C configuration of the femur
  Interventions: Procedure: THA using a short stem

INTERVENTIONS:
Procedure: THA using a short stem — Total Hip Arthroplasty using a collarless, triple-tapered cementless short stem (Optimys, produced by Mathys).

SUMMARY:
Total hip arthroplasty (THA) is a widely accepted procedure for the treatment of end-stage hip osteoarthritis. Neck preserving short stems have gained popularity in recent years, as they aim to preserve proximal femoral bone stock and enable a more physiological load transfer. However, the use of these stems in patients with specific femoral deformities, such as DORR Type C femurs, can present unique challenges. DORR Type C femurs are characterized by decreased cortical bone thickness and increased medullary canal width, which can impact the fit and stability of the femoral stem component. Short stem total hip arthroplasty has emerged as a potential solution for these patients, as it aims to preserve proximal femoral bone stock and improve load transfer to the surrounding bone. This study seeks to investigate the measured subsidence of short stem total hip arthroplasty in patients with DORR Type C femur configuration and the clinical outcomes associated with this approach.

DETAILED DESCRIPTION:
In hip arthroplasty, short stems represent a key advancement in the field of bone-preserving surgical techniques. Due to the relatively rapid establishment of short stems, the data situation is lagging behind in some areas, resulting in uncertainties in the indication in certain cases. One of these cases is proximal femurs with a Dorr type C configuration. This bone characteristic complicates the implantation of stems due to a thin cortical bone and a wide femoral canal and has been shown to lead to an increased complication rate. The aim of this study is to evaluate the clinical and radiological outcome of short stem implantation in Dorr type C femur. The study will include all patients who underwent implantation of the "Optimys" short stem from Mathys between January 1, 2018 and December 31, 2020 at the hospital Ordensklinikum Linz Barmherzige Schwestern. In addition, patients must have a type C femur according to Dorr. During a follow-up period of at least two years, the Harris Hip Score, the UCLA Activity-level Scale and the Singh Index are used to evaluate the clinical course. Radiological evaluation is carried out using pre- and postoperative X-rays, which together enable an EBRA-FCA.

A statement on the migration behavior of the cementless implanted short stem in Dorr type C femur is expected. To date, it has been controversially discussed whether a Dorr type C femur provides enough structural support to achieve good primary stability for a cementless implanted short stem with tapered-wedge design. If this were not the case, the excessive migration behavior would lead to subsidence and subsequently to aseptic stem loosening and even complete failure of the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* THA using Optimys short stem from 1.1.2018 bis 31.12.2020 in the institution.
* Typ C Femur according to Dorr

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 108 patients were eligible, of which 55 underwent routine follow-ups. Complete data was available from 44 patients. 22 patients each were male and female. Mean age at surgery was 68.3 years. Mean BMI was 27.9 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Stem Subsidence | 2 years
  Subsidence of the femoral stem, measured in mm

SECONDARY OUTCOMES:
HHS | 2 years
  Harris Hip Score, 0-100 points. 0 points indicate worst, 100 points indicate best outcome.
OHS | 2 years
  Oxford Hip Score, 0-48points 0 points indicate worst, 48 points indicate best outcome.
SF-12 | 2 years
  Short Form 12, 12 questions with 0-100 points. 0 points indicate worst, 100 points indicate best outcome. Norm-Based-Scoring is used.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordensklinikum Linz Barmherzige Schwestern, Linz, Austria

IPD SHARING:
Plan to Share IPD: Undecided